CLINICAL TRIAL: NCT02812355
Title: High Dose Versus Low Dose Heparinization in Patients Undergoing Offpump Coronary Artery Bypass
Brief Title: Randomized Anticoagulation Trial in Opcab (RATIO)
Acronym: RATIO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Lecco (Other)
Responsible Party: Principal Investigator, Michele Triggiani, MD, PhD, Azienda Ospedaliera di Lecco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT n. 2016-001529-15
Record Dates: First submitted 2016-06-22; First posted 2016-06-24 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Ischemic Heart Disease
Keywords: off-pump; coronary artery bypass; heparinization
MeSH Terms: conditions — Myocardial Ischemia | interventions — Heparin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- half heparinization (Experimental): heparin I.V. 150 U/kg
  Interventions: Drug: Heparin
- full heparinization (300 U/kg) (Active Comparator): heparin I.V. 300 U/kg
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Heparin

SUMMARY:
The RATIO Study is a multicenter, nationwide, randomized, controlled, single blinded, unfunded trial of n. 900 patients undergoing multivessel OPCAB (≥2 grafts). This study is designed to test in patients undergoing off-pump coronary artery bypass surgery the hypothesis that full (high dose, 300 U/kg) and half (low dose,150 U/kg) heparinization are not different in terms of thrombotic complications and major perioperative bleeding events (null hypothesis).

DETAILED DESCRIPTION:
Off-pump coronary artery bypass grafting (OPCAB) is an established alternative to on-pump coronary artery bypass grafting (CABG). OPCAB determines a pro-coagulant state potentially deleterious on grafts patency, that is not counterbalanced by the adverse effects of cardiopulmonary bypass on coagulation occurring in CABG, and that lasts as long as one month. Therefore in OPCAB systemic heparinization is necessary to prevent thrombotic complications during transitory occlusion of coronary arteries and grafts. An internationally accepted standard intra-operative anticoagulation protocol for OPCAB has not yet been defined, and heparinization in OPCAB is a highly variable practice. The intraoperative anticoagulation regimen adopted in patients undergoing OPCAB may influence major postoperative outcomes, such as bleeding, transfusion requirements, inflammatory response, myocardial ischemia and grafts patency, but it has never been the object of large-scale randomized controlled trial (RCT). The 2 most widespread intraoperative anticoagulation protocols in OPCAB are represented by full (300 U/kg) or half (150 U/kg) heparinization, with target ACT ranging from 200 sec to >480 sec.

Patients enrolled in the study will be randomized to receive full or half heparinization in a 1:1 ratio using a randomization schedule blocked by site. Randomization will take place in the operatory room by the anesthesiologist, and will be blinded to the surgeon.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients electively undergoing multivessel OPCAB

Exclusion Criteria:

Acute coronary syndrome, on-going double anti-platelets treatment (the second antiplatelet drug should be suspended 5 days before surgery), on-going intravenous heparin or sub-cutaneous low molecular weight heparin, known coagulopathy, documented liver disease, chronic renal failure (creatinine ≥ 2 mg/dl) or previous renal transplantation surgery, previous cardiac surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Composite vascular | 30 days post-operatively
  Death from vascular causes, perioperative myocardial infarction, stroke.
Composite major bleeding | 48 hours post-operatively
  Redo for excessive bleeding, cardiac tamponade, transfusion ≥3 Units of packed red cells or of platelets.

SECONDARY OUTCOMES:
Post-operative bleeding | 48 hours post-operatively
  Total bleeding evaluated the morning after surgery (ml.)
Transfusion of packed red cells (<3 Units) or of platelets | 30 days post-operatively
Peak value of cardiac biomarker | 30 days post-operatively
Transient ischemic cerebral attack | 30 days post-operatively
Mesenteric ischemia (angiography or CT scan) | 30 days post-operatively
Pulmonary embolus (angiography or CT scan) | 30 days post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Michele NR Triggiani, MD, PhD, Principal Investigator — ASST Lecco
Locations (3):
- Jilin Heart Hospital, Changchun, Jilin, China
- Italy (2):
  - ASST Lecco, Lecco
  - Azienda Ospedaliera Universitaria di Sassari, Sassari

IPD SHARING:
Plan to Share IPD: No